CLINICAL TRIAL: NCT03965754
Title: Assessing the Impact of myHealth Rewards Program-related Email Communications on Enrollment
Brief Title: Assessing the Impact of myHealth Rewards Enrollment Emails
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Other Study IDs: 2019-0404
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Health Promotion; Wellness Programs
Keywords: Prospect theory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No email: No email will be sent out to this subset of GHP members during the week that the other emails are sent.
- Standard email reminder: The standard email reminder mentions the average premium savings, the speed and ease of starting the process, and the deadline for registering and having health measures on file, plus it provides two button links for registering and finding free health screenings where health measures can be collected and registered at one convenient time and location.
  Interventions: Behavioral: Email reminder
- Social norms email: The social norms email notes that a majority (78%) of GHP members' colleagues had enrolled in 2018, it provides a testimonial from a medical director at Geisinger's Commonwealth School of Medicine, stating the ways in which myHealth Rewards helped that doctor personally, and it emphasizes the simplicity and ease of taking the first step toward enrollment.
  Interventions: Behavioral: Social norms; Behavioral: Email reminder
- Loss framing: The loss framing email suggests that GHP members are currently "throwing away" a precise dollar amount (over $2,000) by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action.
  Interventions: Behavioral: Loss framing; Behavioral: Email reminder

INTERVENTIONS:
Behavioral: Social norms — This intervention introduces recipients to descriptive social norms specifying that a majority of their colleagues have signed up for the program, which sets a normative standard against which recipients are expected to compare themselves and to change their behavior accordingly (i.e., when they realize that their behavior is discrepant from that of relevant others). The personal testimonial from a Geisinger medical director serves as a personal exemplar intended to further enhance the effect of the social norms with an implicit indication that the intended behavior is desirable and feasible.
  Other Names: Descriptive norms; Social proof
  Groups: Social norms email
Behavioral: Loss framing — This intervention frames the status quo as a state from which recipients, via inaction, are slated to forfeit a sizable and precise monetary amount to which they should otherwise feel entitled (via loss aversion and the endowment effect). People tend to be risk-seeking in the domain of losses; therefore, this intervention is hypothesized to increase enrollment in the hope of achieving zero loss by meeting program goals, as opposed to a sure loss via inaction.
  Other Names: Endowment effect
  Groups: Loss framing
Behavioral: Email reminder — This intervention is a standard email reminder that mentions the average premium savings, the speed and ease of starting the process, and the deadline for registering and having health measures on file, plus it provides two button links for registering and finding screenings.
  Groups: Loss framing; Social norms email; Standard email reminder

SUMMARY:
The purpose of the study is to evaluate, prospectively, the potential impact of different email message conditions (no email, standard promotional email, social norms, and loss framing) on enrollment in a wellness program (myHealth Rewards) by Geisinger Health Plan (GHP) members.

DETAILED DESCRIPTION:
The myHealth Rewards wellness program managed by GHP rewards those GHP members who carry their insurance through employment at Geisinger with reduced health insurance premiums over the course of the following year, if members register for the program and have their health measures on file by the enrollment deadline and are then able to meet their health goals by the respective due date. In spite of the potential savings to health plan members and the wellness program's potential to motivate engagement in healthy activities (with consequent improvement in health outcomes), over 20% of eligible GHP members have not yet enrolled in 2019, even after receiving promotional email communications and reminders. Therefore, the current study was developed to test whether different versions of emails are more effective than a standard reminder email or no-email condition in increasing myHealth Rewards login and enrollment rates. The standard email reminder mentions the average premium savings, the ease of the registration process, and the deadline for registering and having health measures on file, plus it provides links for registering and finding free health screenings where health measures can be collected and registered at one convenient time and location. The social norms email notes that a majority (78%) of GHP members' colleagues had enrolled in 2018, it provides a testimonial from a medical director at Geisinger's Commonwealth School of Medicine, stating the ways in which myHealth Rewards helped that doctor personally, and it emphasizes the simplicity and ease of taking the first step toward enrollment. The loss framing email suggests that GHP members are currently "throwing away" a precise monetary amount in savings by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action. It is hypothesized that, on average, each of the emails will increase enrollment compared with no email. Among GHP members who never enrolled in the past, it is hypothesized that the standard email reminder will not be as effective as the social norms and loss framing emails. Therefore, email conditions will be compared separately among those who did and did not register in 2018. Findings will help inform how best to increase enrollment in a wellness program among health plan members who have already received past promotional communications and who may or may not have participated in the past.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger employees who are benefits subscribers

Exclusion Criteria:

* Those who had already registered for myHealth Rewards in 2019, up through May 6, 2019
* New Geisinger employees hired between December 1, 2018 and May 6, 2019
* Existing Geisinger employees who transitioned from non-subscribers in 2018 to subscribers in 2019

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population consists of Geisinger Health Plan members who are benefits subscribers.
Sampling Method: Probability Sample
Enrollment: 5697 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Email | Standard Email Reminder | Social Norms Email | Loss Framing
Started (No email bounce information was available, so this number includes all people emailed.) | 1422 | 1425 | 1425 | 1425
Completed (Given no bounce information, all emails were considered received, which we counted as completion.) | 1422 | 1425 | 1425 | 1425
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline outcome measure was not applicable, since enrollment and login in response to the email was the outcome. There was no previous email, and participants were selected for not having enrolled in the year of the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Email | Standard Email Reminder | Social Norms Email | Loss Framing | Total
Number analyzed (Participants) | 1422 | 1425 | 1425 | 1425 | 5697
Age, Categorical [Count of Participants; unit: Participants] — Only de-identified data on email engagement was collected; no age data was collected.
  Participants
    <=18 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    >=65 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — Only de-identified data on email engagement was collected; no sex or gender data was collected.
  Participants
    Female | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1422 | 1425 | 1425 | 1425 | 5697

OUTCOME MEASURES:

1. Primary Outcome: Enrollment (7 Days)
Description: Enrollment in the myHealth Rewards program (yes/no) within 7 full days of the beginning of the intervention (i.e., when the emails are first sent).
Time Frame: 7 days, from May 7 through 13, 2019
Population: We planned a priori to specifically compare the conditions within two groups: employees who previously enrolled and employees who never enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | No Email | Standard Email Reminder | Social Norms Email | Loss Framing
Number analyzed (Participants) | 1422 | 1425 | 1425 | 1425
Participants
  Previously Enrolled: number analyzed (Participants) | 741 | 742 | 742 | 742
  Previously Enrolled | 29 | 126 | 88 | 145
  Never Enrolled: number analyzed (Participants) | 681 | 683 | 683 | 683
  Never Enrolled | 4 | 8 | 6 | 13
Statistical Analysis 1: Comparison: No Email vs Loss Framing; We conducted a logistic regression with the three email conditions as dummy variables with no email as the reference group (among employees who previously enrolled in the program); Test type: Superiority; p < .001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 5.96, 95% CI 2-sided [4.00 to 9.18]
Statistical Analysis 2: Comparison: No Email vs Standard Email Reminder; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 5.02, 95% CI 2-sided [3.36 to 7.76]
Statistical Analysis 3: Comparison: No Email vs Social Norms Email; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 3.30, 95% CI 2-sided [2.17 to 5.17]
Statistical Analysis 4: Comparison: No Email vs Loss Framing; We conducted a logistic regression with the three email conditions as dummy variables with no email as the reference group (among employees who never enrolled in the program); Test type: Superiority; p = .038, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.16 to 11.71]
Statistical Analysis 5: Comparison: No Email vs Standard Email Reminder; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = .256, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.63 to 7.54]
Statistical Analysis 6: Comparison: No Email vs Social Norms Email; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = .531, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.43 to 5.89]
Statistical Analysis 7: Comparison: Standard Email Reminder vs Loss Framing; We conducted a logistic regression with the two experimental conditions as dummy variables with the standard email as the reference group (among employees who previously enrolled in the program); Test type: Superiority; p = .202, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.91 to 1.54]
Statistical Analysis 8: Comparison: Standard Email Reminder vs Social Norms Email; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = .005, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.49 to 0.88]
Statistical Analysis 9: Comparison: Standard Email Reminder vs Loss Framing; We conducted a logistic regression with the two experimental conditions as dummy variables with the standard email as the reference group (among employees who never enrolled in the program); Test type: Superiority; p = .276, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.69 to 4.16]
Statistical Analysis 10: Comparison: Standard Email Reminder vs Social Norms Email; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = .592, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.25 to 2.16]

2. Primary Outcome: Logging in (7 Days)
Description: Logging into the myHealth Rewards program (yes/no) within 7 full days of the beginning of the intervention.
Time Frame: 7 days, from May 7 through 13, 2019
Population: There was no login data for participants in the "No email" group, as the website link was provided by the email. In addition, we planned a priori to specifically compare the conditions within two groups: employees who previously enrolled and employees who never enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | No Email | Standard Email Reminder | Social Norms Email | Loss Framing
Number analyzed (Participants) | 0 | 1425 | 1425 | 1425
Participants
  Previously Enrolled: number analyzed (Participants) | 0 | 742 | 742 | 742
  Previously Enrolled | 0 | 182 | 117 | 222
  Never Enrolled: number analyzed (Participants) | 0 | 683 | 683 | 683
  Never Enrolled | 0 | 25 | 19 | 42
Statistical Analysis 1: Comparison: Standard Email Reminder vs Loss Framing; Test type: Superiority — We conducted a logistic regression with the two experimental conditions as dummy variables with the standard email as the reference group (among employees who previously enrolled); p = .020, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.04 to 1.65]
Statistical Analysis 2: Comparison: Standard Email Reminder vs Social Norms Email; We conducted a logistic regression with the two experimental conditions as dummy variables with the standard email as the reference group (among employees who previously enrolled); Test type: Superiority; p < .001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.44 to 0.75]
Statistical Analysis 3: Comparison: Standard Email Reminder vs Loss Framing; We conducted a logistic regression with the two experimental conditions as dummy variables with the standard email as the reference group (among employees who never enrolled); Test type: Superiority; p = .359, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.41 to 1.38]
Statistical Analysis 4: Comparison: Standard Email Reminder vs Social Norms Email; Test type: Superiority — We conducted a logistic regression with the two experimental conditions as dummy variables with the standard email as the reference group (among employees who never enrolled); p = .035, Regression, Logistic; We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.05 to 2.90]

ADVERSE EVENTS:
Time Frame: No adverse events were evaluated.
Description: We only received aggregate information about email engagement with no individual-level information collected (including those for adverse events).
Arm/Group | No Email | Standard Email Reminder | Social Norms Email | Loss Framing
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
For this study, we only received data about engagement with the email. Individual patients were not identified and demographic information such as age, sex, or gender were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT03965754/Prot_SAP_000.pdf